CLINICAL TRIAL: NCT02330068
Title: Microbiome of Depression &Amp; Treatment Response to Citalopram: A Feasibility Study
Brief Title: Microbiome of Depression & Treatment Response to Citalopram
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, William V. Bobo, M.D., PI, Mayo Clinic
Other Study IDs: 14-002154
Record Dates: First submitted 2014-12-09; First posted 2015-01-01 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2017-12

CONDITIONS: Major Depressive Disorder, Bipolar I and Bipolar II
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Citalopram

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, saliva and stool samples will be collected at three time points.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Controls: Males and females ages 18-55 without Major Depressive Disorder, Bipolar I or Bipolar II who are not on an antidepressant and do not have a first degree relative with a diagnosis of Major Depressive Disorder and not currently taking citalopram.
- Cases: Male or female participants ages 18-55 with Major Depressive Disorder, Bipolar I or Bipolar II whom antidepressant treatment is deemed necessary will be given citalopram.
  Interventions: Drug: citalopram

INTERVENTIONS:
Drug: citalopram — Cases
  Other Names: Celexa
  Groups: Cases

SUMMARY:
The purpose of this study is to evaluate the feasibility of developing a microbiome probe of depression and to evaluate the microbiome change in a preliminary analysis of treatment response (n=20) vs. non response (n=20) to the antidepressant citalopram. This study is a 12 week open trial that will enroll approximately 80 participants (anticipated 40 study completers with paired biomarker data) with an episode of major depression, Bipolar I or Bipolar II and 40 age- and sex-matched healthy controls.

DETAILED DESCRIPTION:
The study will be conducted at Mayo Clinic Jacksonville Department of Psychiatry (recruit up to 10 patients and 10 controls with paired data) and Mayo Clinic Depression Center in Rochester (recruit up to 30 patients and 30 controls with paired data). Patients with major depression, Bipolar Disorder I or Bipolar Disorder II confirmed by structured diagnostic interview (SCID) and moderate symptom severity (Quick Inventory of Depressive Symptomatology or S-C16) will be enrolled in the 12 week study. We will explore the gut microbiome (and its genetic material) and gut-brain markers of inflammation (cortisol, cytokines) from stool specimens and serum samples, respectively. Collections will be at baseline, week 2, and week 12 of the study. Healthy controls matched for age, sex (including menopausal status of female subjects), and body-mass index (BMI) will have only baseline stool and serum collections. Statistical t-tests will be used to assess baseline differences between patient and controls in microbiome and inflammatory markers. Treatment response (50% reduction in QIDS), treatment remission (QIDS-C16 < 6) will be analyzed with change in microbiome and inflammation markers. Correlational analysis with multiple testing corrections will be conducted between depression symptom severity and measures of cortisol, cytokines, and gut microbiome composition.

This study will focus on early translation of Dr. Fryer and Dr. Chia's research and will bring the gut-brain interface to the field of individualizing treatment to patients who struggle with depression. This project will provide insight into how gut microbiota may be implicated in depression, how antidepressant treatments alter microbiota composition, and how these factors impact key physiologic mediators of depression (i.e. cortisol and cytokine levels). The public health implications of more focused drug development and treatment for depression are substantial.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients or inpatients with nonpsychotic major depressive disorder (MDD) or Bipolar I or II Disorder.
* A score of >16 on the QIDS
* Outpatients or inpatients for whom antidepressant treatment is deemed appropriate by the treating clinician
* Subjects who are between 18-55 years of age

Exclusion Criteria:

* Contraindications to citalopram treatment
* Axis I or II disorder other than depression that is the primary reason for seeking treatment intervention and/or psychiatric care
* Subjects diagnosed with Borderline Personality Disorder (BPD) as their primary diagnosis.
* For healthy controls, a first degree relative who has been diagnosed with an Axis I disorder
* Patients with schizophrenia, schizoaffective disorder, or bipolar I disorder
* Antidepressant treatment within 4 days of study (1 week if fluoxetine). Subjects currently on antidepressant medication with subtherapeutic results in terms of depression management after providing informed consent, will undergo a medication taper and discontinuation prior to initiation of citalopram treatment. The subject must be off of previous antidepressants for at least 4 days week prior to starting citalopram (1 week if fluoxetine). The subject will be closely monitored by the research study psychiatrist (with or without additional monitoring from primary clinical psychiatric providers). The medication taper is left up to the research study psychiatrist in consultation with patient's primary care or psychiatric provider. Study subjects who cannot be safely tapered from their medication or experience adverse effects during the taper will be excluded from the study
* Study subjects using their antidepressant medication for management of nicotine dependence, chronic pain, migraine prophylaxis, or other diagnoses will not be eligible for the study unless they remain on a stable dose of the medication for the 12 weeks of the study.
* Trazodone, melatonin, and diphenhydramine may be used as rescue medications for insomnia. Benzodiazepines may be used for treatment of anxiety, not to exceed 4 mg/24 hour of lorazepam
* Subjects who are currently on an antibiotic or an antibiotic within 2 weeks. (Topical antibiotics are OK)
* Daily use of aspirin, NSAID's or Warfarin (low dose of baby aspirin OK)
* Subjects unable to give informed consent are excluded
* Pregnant subjects will be excluded
* Subjects who are currently breastfeeding and who plan to continue breastfeeding will be excluded
* Postmenopausal women are not eligible for this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The investigators will enroll 80 participants, both male and female with the goal of having 20 paired data of responders and 20 non-responders each. Forty age-matched healthy controls will also be recruited. The investigators will recruit 100 subjects anticipating drop outs or inability to participate fully with microbiome sample collection and /or at least paired biological specimens before and after treatment. The Mayo Clinic Jacksonville patients (n=10) will be matched with Mayo Clinic Jacksonville controls (n=10) and the Mayo Clinic Rochester patients (n=30) will be matched with the Mayo Clinic Rochester controls (n=30).
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The potential differences in the microbiome between depressed patients and healthy controls | Over 12 weeks
  The gut microbiome of depressed patients is different from that of age-, sex-, menopause-, and BMI-matched healthy controls

SECONDARY OUTCOMES:
Microbiome change in treatment response vs. non-response to citalopram | Over 12 weeks
  The gut microbiome change of patients that respond to citalopram is different
Inflammatory markers of depression and their relationship to the microbiome | Over 12 weeks
  Changes in inflammatory markers of depression correspond to changes in depression symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: William Bobo, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota